CLINICAL TRIAL: NCT00247624
Title: Hypnotics in the Treatment of Psychiatric Disorders
Brief Title: Improving Sleep and Psychological Functioning in People With Depression and Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Sumitomo Pharma America, Inc. (Industry); Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R34MH070821 (NIH); DSIR 83-ATSO; R34MH070821 (NIH)
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Sleep Initiation and Maintenance Disorders; Depression
Keywords: Depression; Hypnotics; Sleep; Quality of Life; Insomnia; Suicide
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Suicide | interventions — Eszopiclone; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Participants will receive treatment with eszopiclone and fluoxetine
  Interventions: Drug: Eszopiclone; Drug: Fluoxetine
- B (Active Comparator): Participants will receive treatment with placebo and fluoxetine
  Interventions: Drug: Fluoxetine; Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone — Eszopiclone 3 mg every night for 8 weeks
  Arms: A
Drug: Fluoxetine — Fluoxetine 20 mg every morning for 9 weeks
Drug: Placebo — Placebo every night for 8 weeks
  Arms: B

SUMMARY:
This study will evaluate the safety and effectiveness of treatment with both a sleeping pill and antidepressant medication in improving sleep and psychological functioning in people with depression and insomnia.

DETAILED DESCRIPTION:
Chronic insomnia is one of the most common symptoms that individuals experience during a major depressive episode. Insomnia may lead to increased risk for recurrence of major depression, as well as poor quality of life and increased risk of suicide. Studies have shown that treating insomnia during a major depressive episode may not only help reduce symptoms of major depression during the day, but also improve an individual's general quality of life. Thus, sleeping pills, also known as hypnotics, are commonly prescribed for people with psychiatric disorders. However, little is known about the safety and efficacy of combining sleeping pills with antidepressant medications. This study will evaluate the safety and effectiveness of treatment with both a sleeping pill and antidepressant medication in improving sleep and psychological functioning in people with depression and insomnia.

Participants in this double-blind study will first receive fluoxetine, an antidepressant medication, for 1 week. Participants whose symptoms of insomnia subside after this initial week will continue on fluoxetine for the duration of the study and will not receive sleeping pills. Those who do not experience an improvement in their symptoms of insomnia after 1 week will be randomly assigned to receive either placebo or eszopiclone, which is a sleeping pill, in addition to fluoxetine. All treatments will be given for 8 weeks. Participants will attend study visits at various points throughout the treatment phase. Follow up visits will occur periodically over the next 4 months. Assessments will include physiological measures during sleep, mood, suicidal thinking, quality of life and actigraphy, which measures the amount of movement during sleep.

ELIGIBILITY:
Inclusion Criteria:

* Score of greater than 10 on the Primary Care Evaluation of Mental Disorders Patient Health Questionnaire (PRIME-MD-PHQ) telephone screen
* Diagnosis of major depressive episode based on the Structured Clinical Interview for DSM-IV (SCID)
* Score of greater than 20 on the Hamilton Rating Scale for Depression
* Meets research diagnostic criteria for insomnia disorder at least 4 nights per week
* Reported mean sleep latency greater than 30 minutes and mean sleep efficiency less than 85%
* Suitable for outpatient treatment

Exclusion Criteria:

* Use of any psychotropic medications within 2 weeks of initial screening
* Bipolar disorder, schizophrenia, psychotic depression, or any other psychotic disorder
* Uncontrolled asthma or chronic obstructive pulmonary disease
* Chronic pain that may be a significant sleep-disturbing factor
* Uncontrolled thyroid disease
* Poorly controlled diabetes mellitus
* Poorly compensated congestive heart failure
* Currently taking lipophilic beta blockers, opioids, glucocorticoids, theophylline, or other medications known to interfere with sleep
* History of intolerance or treatment resistance to either fluoxetine or eszopiclone
* Inability to abstain from taking any psychotropics other than the study medications during the course of the protocol, including sedating antihistamines
* Use of any herbal or naturopathic treatments for sleep or mood (i.e., St. John's wort, melatonin, kava kava, valerian root, etc.)
* Currently undergoing behavioral, cognitive-behavioral, or interpersonal therapy
* Pregnant or breastfeeding
* Agrees to use an effective form of contraception for the duration of the study
* Uncontrolled symptoms of menopause, including hot flashes
* Uncontrolled hypertension (systolic blood pressure consistently greater than 140 mm Hg, diastolic blood pressure consistently greater than 90 mm Hg)
* Diagnosis of sleep apnea, periodic limb movement disorder, or restless leg syndrome
* Reports habitual bedtime earlier than 9 PM or later than 1 AM more than 2 times per week
* Reports habitual rising time later than 9 AM more than 2 times per week
* Body mass index greater than 30
* Consumes more than 3 alcoholic beverages per day
* Consumes more than 4 caffeinated beverages per day
* Habitual smoking between 11 PM and 7 AM
* Use of illicit drugs
* Score greater than 24 on the Mini Mental State Examination
* Determined to be incompetent
* Determined to be at imminent risk for suicide
* More than 5 lifetime SCID diagnoses of major depressive episodes
* More than 3 failed antidepressant trials during the current episode of depression, as determined by the Antidepressant Treatment History Form
* A course of electroconvulsive therapy during the present depressive episode

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-10; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W. Vaughn McCall, MD, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences; Department of Psychiatry and Behavioral Medicine, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] McCall WV, Reboussin BA, Cohen W. Subjective measurement of insomnia and quality of life in depressed inpatients. J Sleep Res. 2000 Mar;9(1):43-8. doi: 10.1046/j.1365-2869.2000.00186.x. PMID 10733688
- [Background] Zammit GK, Weiner J, Damato N, Sillup GP, McMillan CA. Quality of life in people with insomnia. Sleep. 1999 May 1;22 Suppl 2:S379-85. PMID 10394611
- [Derived] McCall C, McCall WV. Objective vs. subjective measurements of sleep in depressed insomniacs: first night effect or reverse first night effect? J Clin Sleep Med. 2012 Feb 15;8(1):59-65. doi: 10.5664/jcsm.1664. PMID 22334811
- [Derived] McCall WV, D'Agostino R Jr, Rosenquist PB, Kimball J, Boggs N, Lasater B, Blocker J. Dissection of the factors driving the placebo effect in hypnotic treatment of depressed insomniacs. Sleep Med. 2011 Jun;12(6):557-64. doi: 10.1016/j.sleep.2011.03.008. Epub 2011 May 20. PMID 21601519
- [Derived] McCall C, McCall WV. Comparison of actigraphy with polysomnography and sleep logs in depressed insomniacs. J Sleep Res. 2012 Feb;21(1):122-7. doi: 10.1111/j.1365-2869.2011.00917.x. Epub 2011 Mar 29. PMID 21447050
- [Derived] McCall WV, Blocker JN, D'Agostino R Jr, Kimball J, Boggs N, Lasater B, Haskett R, Krystal A, McDonald WM, Rosenquist PB. Treatment of insomnia in depressed insomniacs: effects on health-related quality of life, objective and self-reported sleep, and depression. J Clin Sleep Med. 2010 Aug 15;6(4):322-9. PMID 20726279
- [Derived] McCall WV, Blocker JN, D'Agostino R Jr, Kimball J, Boggs N, Lasater B, Rosenquist PB. Insomnia severity is an indicator of suicidal ideation during a depression clinical trial. Sleep Med. 2010 Oct;11(9):822-7. doi: 10.1016/j.sleep.2010.04.004. Epub 2010 May 15. PMID 20478741

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluoxetine (FLX) Plus Eszopiclone (ESZ): Participants will receive treatment with eszopiclone and fluoxetine
- FLX Plus Placebo: Participants will receive treatment with placebo and fluoxetine
Period: Overall Study
Arm/Group | Fluoxetine (FLX) Plus Eszopiclone (ESZ) | FLX Plus Placebo
Started | 30 | 30
Completed | 25 | 26
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoxetine (FLX) Plus Eszopiclone (ESZ) | FLX Plus Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (11.7) | 38.0 (12.5) | 41.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 10 | 10 | 20
BASIS 32 DLRF [Mean (Standard Deviation); unit: units] — The BASIS 32 psychometric includes several subscales, including "daily living and role functioning" (DLRF). This subscale is rated from 0-4, with higher scores indicating a greater deal of difficulty in this dimension
  units | 1.9 (0.7) | 2.0 (0.7) | 2.0 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Daily Living and Role Functioning (DLRF) Basis-32 Subscale Ratings
Description: The BASIS 32 psychometric includes several subscales, including "daily living and role functioning" (DLRF). These subscales are rated from 0-4, with higher scores indicating a greater deal of difficulty in this dimension and lower scores denoting better outcomes. Measured weekly for 9 weeks. Reported as mean of 9 weeks.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluoxetine (FLX) Plus Eszopiclone (ESZ) | FLX Plus Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 0.81 (0.64) | 1.2 (0.72)

2. Primary Outcome: Relation to Self/Others (RSO) Basis-32 Subscale Ratings
Description: The BASIS 32 psychometric includes several subscales, including "relation to self and others" (RSO). These subscales are rated from 0-4, with higher scores indicating a greater deal of difficulty in this dimension. Measured weekly for 9 weeks. Reported as mean of 9 weeks.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluoxetine (FLX) Plus Eszopiclone (ESZ) | FLX Plus Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 0.74 (0.71) | 1.04 (0.77)

3. Primary Outcome: Quality of Life Ratings, as Measured by the Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q)
Description: The Q-LES-Q is scored from 0-100, with higher scores better than lower. Measured weekly for 9 weeks. Reported as mean of 9 weeks.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluoxetine (FLX) Plus Eszopiclone (ESZ) | FLX Plus Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 50.2 (8.11) | 46.9 (9.0)

4. Secondary Outcome: Insomnia Severity Index (ISI)
Description: The Insomnia Severity Index has seven questions. The seven answers are added up to get a total score, range 0-28. Lower scores represent better outcomes. Total score categories: 0-7 = No clinically significant insomnia, 8-14 = Subthreshold insomnia, 15-21 = Clinical insomnia (moderate severity), 22-28 = Clinical insomnia (severe).
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluoxetine (FLX) Plus Eszopiclone (ESZ) | FLX Plus Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 21.1 (4) | 20.2 (4.1)

ADVERSE EVENTS:
Arm/Group | Fluoxetine (FLX) Plus Eszopiclone (ESZ) | FLX Plus Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes